CLINICAL TRIAL: NCT02213614
Title: Lithium Water Use in Gun Violence Prevention
Brief Title: Lithium Water in Gun Violence Prevention
Acronym: LWGVP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: American Society Of Thermalism And Climatology Inc (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: vio829429989
Record Dates: First submitted 2014-08-05; First posted 2014-08-11 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2015-06

CONDITIONS: Assault by Handgun Discharge; Violence; Homicide; Sexual Assault by Bodily Force; Substance Abuse Problem
MeSH Terms: conditions — Substance-Related Disorders | interventions — Natural Childbirth

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Spring Lithium Water (Experimental): The Long term goal of this research project is the implementation of an effective, inexpensive therapy in communities with high risk of violence. Therapy will be based on a daily dietary supplement LIWA at appropriate doses.
  The short-term objective is to prove that Lithium water (LIWA) as a daily supplement is an intervention that prevents gun violence from occurring, and is a factor that decrease the violence for gun in our communities Gun violence poses a serious threat to America's children and youth. Existing data clearly point to the need for improved strategies for keeping guns out of the hands of children and youth and those who would harm them.
  Interventions: Dietary Supplement: Lithium Water
- Placebo: Natural Spring water (Experimental): This group will be drink natural spring water for 4 months in tres cicles
  Interventions: Dietary Supplement: placebo: spring mineral water; Other: natural spring water

INTERVENTIONS:
Dietary Supplement: Lithium Water — Supply daily doses of Lithium water in form bottled mineral water
  Other Names: Spring mineral water; Crazy water
  Arms: Spring Lithium Water
Dietary Supplement: placebo: spring mineral water — Drink spring natural water a placebo 3 times a day
  Other Names: natural water; spring water
  Arms: Placebo: Natural Spring water
Other: natural spring water — A group will drink natural spring water for 4 months
  Other Names: natural water; spring water
  Arms: Placebo: Natural Spring water

SUMMARY:
The word lithium frequently conjures images of catatonic psychiatric patients and side effects so severe that premature death is commonplace. But naturally occurring lithium is a far cry from pharmaceutical grades. Found in the soil, water and certain foods, it is an essential mineral for maintaining physical and mental health. When exposure is low, suicide rates, mental illness and violent crime increase

DETAILED DESCRIPTION:
Lithium has a long history of use in the treatment of mental disorders. However, it hasn't been until recently that scientists began exploring the psychiatric implications of naturally occurring lithium in the water supply.

As stated in the article, Foods Rich in Lithium And Lithium Supplements:

"Research suggests that locations with the highest concentration of lithium tend to have the lowest rates of depression and violent crime. These studies have been conducted across the globe in different climates with different natural habits and diets. Researchers have therefore concluded that this phenomenon is fairly universal."

A study in the United States agrees with these findings. According to Everything Addiction:

"In a 1990 study of 27 Texas counties, researchers found an "inverse association of tap water lithium content in areas of Texas with the rates of mental hospital admissions, suicides, homicides, and certain other crimes." It was also discovered that young men incarcerated for violent crimes in some parts of Texas had disproportionately low lithium levels. Schrauzer and Shrestha discovered that the negative correlation was confirmed," especially in the south-central region of the state where high suicide mortality rates correspond to low lithium concentrations."'

Another study published in the British Journal of Psychiatry had similar results. Researchers at Oita University examined the suicide rates in Japan's Oita prefecture. The team discovered that cities with higher levels of natural lithium in the public water supply had lower rates of suicide overall.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 14-60.
* Existence of alcoholism, substance abuse, violence antecedent, suicide history Answered all questions in the pre-treatment safety questionnaire. Gave their oral and written consent to participate in the trial.

Exclusion Criteria:

Patients with renal failure, cardiovascular insufficiency, Addison's disease and untreated hypothyroidism.

Pregnancy. Patients who have vomiting or diarrhea or if fluid or salt (sodium) intake is increased or decreased.

Inadequate communication with examiner. Participation in another clinical study, either concurrent with this trial or in the 3 months preceding it.

Inability to sign a consent form.

Ages: 14 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 400 (Estimated)
Dates: Start 2014-08; Primary Completion 2015-12 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Change behavioral tendencies due to lithium water treatment | 1 year
  During the next study we will analyze the behavior of violent tendencies in three counties of New Jersey (ESSEX, Hudson and Passaic) during the years 2010-2013, different parameters were identified such as:
  Firearms violence Domestic violence Killings Rape Theft Suicides Alcoholism Substance abuse We will Identify 400 individuals randomly with one or more of these known behaviors, which are invited to participate in the study, we will administer them a psycho-social test, a history clinical psycho-social study, levels of lithium in blood test and associated general tests, in addition to EEG, and neuro-physiological studies.
  500 mcg will be given to one group which will indicate them a daily supplement of lithium water while the other group will only receive mineral spring water as a placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Garis Silega, Principal Investigator — American Society of Thermalism and Climatology; Garis Silega, Doctor, Study Director — American Society of Thermalism and Climatology
Locations (1):
- Gaviota Clinic, Newark, New Jersey, United States